CLINICAL TRIAL: NCT04168151
Title: Efficacy of Trans Alveolar Pressure Measurement as an Index for Lung Recruitment in Post Cardiac Surgery Hypoxic Patients.
Brief Title: Trans Alveolar Pressure Measurement as an Index for Lung Recruitment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ibrahim Mabrouk Ibrahim, assistant lecturer of anesthesia, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Hypoxia
Keywords: post cardiac surgery,; lung recruitment; trans alveolar pressure
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypoxic group (Experimental): hypoxic patients (hypoxic index less than 250)
  Interventions: Other: lung recruitment protocol

INTERVENTIONS:
Other: lung recruitment protocol — lung recruitment protocol applied to postcardiac surgery hypoxic adult patients with measurement of trans alveolar pressure as an index for lung recruitment

SUMMARY:
the study is conducted on hypoxic adult patients underwent open heart surgery after arrival to the intensive care unit and stabilization of patients' hemodynamics to assess the efficacy of transalveolar pressure measurement as an index for lung recruitment.

DETAILED DESCRIPTION:
After one hour from the patient's ICU admission and after stabilization of the patient's haemodynamics, alveolar recruitment will be done for hypoxic patients with hypoxic index less than 250.

The recruitment will be started in the adaptive ventilation mode (AVM mode) using modified stepwise staircase recruitment maneuver in which every 2 minutes positive end-expiratory pressure (PEEP) is increased in increments of 2 cmH2O and the driving pressure will be regulated by AVM mode.

The increase in PEEP will be guided by improvement of dynamic compliance, oxygen saturation and transalveolar pressure (PTA) till near overdistention.

Overdistension will be detected if there are decrease in the mean arterial pressure 25% from the base line value reported after stabilization of the patient's haemodynamics, or decreased oxygen saturation or sudden decrease in dynamic compliance, or inspiratory PTA more than15 cm H2O.

Then PEEP is decreased 2 cm H2O every 3 minutes till a decrease expiratory PTA less than 1 cm H2O, or a decrease in dynamic compliance or a decrease in oxygen saturation ≥ 1% from maximum oxygen saturation is observed (the derecruitment point) then return to a PEEP level 2 cm H2O above the derecruitment point (the optimal PEEP).

Alveolar recruitment will be done once.

ELIGIBILITY:
Inclusion Criteria:

* post cardiac surgery hypoxic adult patients

Exclusion Criteria:

1. Patients with contraindications for the use of esophageal catheter including esophageal ulcerations, tumors, diverticulitis, bleeding varices, recent esophageal or gastric surgery, sinusitis, epistaxis and recent nasopharyngeal surgery.
2. Postoperative severe haemodynamic instability on high inotropic support.
3. Ejection fraction less than 35%.
4. Severe restrictive or obstructive lung disease.
5. Extremes of age (<19 and > 75 years).
6. Morbid obese patients with BMI > 40kg/m2.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
transalveolar pressure | 1 day
  cmH2O
hypoxic index | 1 day

SECONDARY OUTCOMES:
dynamic compliance | 1 day
  ml/cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Mabrouk, Principal Investigator — University of Alexandria; Ahmed Y Ali, MD, Study Director — University of Alexandria; Amal M Ahmed, MD, Study Director — University of Alexandria
Locations (1):
- Alexandria main university hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No